CLINICAL TRIAL: NCT01821664
Title: Vascular Graft Infections - Epidemiology, Best Treatment Options, Imaging Modalities and Impact of Negative Pressure Wound Therapy
Brief Title: Vascular Graft Infections
Acronym: VASGRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2012-0583
Record Dates: First submitted 2013-03-07; First posted 2013-04-01 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Prosthetic Vascular Graft Infection
Keywords: Prosthetic vascular graft infection; negative pressure wound therapy; microbiology; antimicrobial therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (1):
- Prosthetic vascular graft implantation, follow up
  Interventions: Device: Prosthetic vascular graft

INTERVENTIONS:
Device: Prosthetic vascular graft — Implantation of a prosthetic vascular graft
  Other Names: Valsalva Graft, Gelwave TM; Subclavia Graft, Gelwave TM; Longer Ante-Flo Offset branch, Gelwave TM; Lupiae Branched Graft, Gelwave TM; 4 Branched Plexus, Gelwave TM; Bifurcate, Gelwave TM soft; Subclavia Graft straight, Gelwave TM soft; Intergard woven straight, Intervascular "Maquet Getinge Group"; Intergard woven hemabridge, Intervascular "Maquet Getinge Group"; Intergard woven Aortic Arch, Intervascular "Maquet Getinge Group"; Intergard Silver Knitted Bifurcation, Intervascular "Maquet Getinge Group"; Intergard Silver Knitted Straight, Intervascular "Maquet Getinge Group"; InterGard TM knitted Bifurcation, Intervascular "Maquet Getinge Group"; FlowLine Bipore r Heparin ePTFE Vascular Graft, Jotec r GmbH; ePTFE Vascular Graft Regular Wall flex, IMPRA r; ePTFE Vascular Graft Thin Wall flex, IMPRA r; ePTFE Vascular Graft Regular Wall straight, IMPRA r; Gore-Tex Stretch Vascular Graft standard Wall Eptfe, W.L. Gore & Associates, Inl

SUMMARY:
Background: Vascular grafts are increasingly implanted due to an increasing prevalence of atherosclerosis and diabetes, and about 1-6% of vascular procedures are complicated by infection. Mortality attributable to prosthetic vascular graft infections (PVGI) is high. However, there are almost no data regarding best treatment options of such complicated infections. Most recommendations are based on expert opinion and not on clinical trials or cohort observational data analyses. Evaluating infectious and other complications after vascular surgery procedures are important, and additionally, such studies may offer insights for quality improvement and improved patient outcomes. With the first aim investigators will establish an infrastructure for studying PVGI in Zurich. Investigators will take advantage of the Swissvasc registry, a central registry which collects preoperative, operative and discharge data regarding the index vascular surgical interventions. They will create a prospective observational cohort database of all patients who receive a vascular graft (peripheral, aortic, vein) at the University hospital of Zurich (VASGRA Cohort A). Patients with a PVGI will be included in VASGRA Cohort B and followed up using a flow chart with a focus on the course of this infectious complication. Additionally, investigators will establish a biobank with the collection of tissue- and blood samples of patients with PVGI. With the second aim researchers will investigate different diagnostic, clinical and therapeutic research questions nested in the VASGRA Cohort. Firstly, they will address epidemiological questions, such as: determine the incidence and outcome of complications after vascular graft placement; determine risk factors, best treatment strategies and outcome of PVGI, and determine the influence of different antibiotic regimens on the outcome of PVGI due to different bacterial pathogens. Secondly, investigators will determine the accuracy of different imaging techniques (PET/CT and MRI) for the diagnosis of PVGI, and their individual role for the assessment of treatment response. Thirdly, investigators will evaluate the bacterial diversity of vascular wound infections using 16s r-Ribonucleic acid (RNA)amplification, and investigators will explore whether this bacterial diversity does predict disease progression. Here, investigators will also study the impact of negative pressure wound therapy (NPWT) on bacterial diversity in the treatment course of PVGI. Fourthly, investigators will look for cut-off levels of relevant blood leucocytes count, C-reactive protein and procalcitonin raising suspicion of a PVGI. Lastly, investigators will look at histopathological features of excised vascular grafts. Expected value of the project: Results from the proposed study are an important contribution to the field, based on the large sample size, longitudinal design and by unifying clinical and epidemiological science. The very well characterized patient groups and the close connection between vascular surgeons, infectious disease specialists, specialists in nuclear medicine and microbiologist will help to investigate PVGI in depths. Investigators hope to be able to develop guidelines regarding best diagnostic modalities and treatment options in case of vascular graft infections. In the future we plan to examine bacteria retrieved from the PVGI in the laboratory in detail. The recovered bacteria will be examined for antimicrobial susceptibility and their capability to form biofilms. Furthermore investigators will examine how bacterial recovery form explanted grafts could be optimized.

ELIGIBILITY:
Inclusion criteria:

Control patients:

- Vascular graft surgery (peripheral, aortic, vein)

Case patients:

* Patients with previous primary implantation of an aortic or peripheral vascular implant and suspicion of PVGI
* Age >18 years
* Written informed consent

Exclusion criteria:

* Drug or alcohol abuse
* Involvement in a conflicting clinical trial (investigational drug)
* Inability to follow the procedures of the cohort, e.g. due to language problems, psychological disorders or dementia of the subject
* Known or suspected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a vascular surgery at the University hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2013-05; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Vascular graft infection | within 10 years
  Persons are followed up after vascular graft surgery.

SECONDARY OUTCOMES:
Bleeding | 10 years
Foreign body reaction | 10 years
All cause- mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hasse, MD, Principal Investigator — University Hospital Zurich, Div of Infectious Diseases and Hospital Epidemiology
Locations (1):
- University Hospital Zurich, Div of Infectious Diseases and Hospital Epidemiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Husmann L, Huellner MW, Ledergerber B, Anagnostopoulos A, Stolzmann P, Sah BR, Burger IA, Rancic Z, Hasse B; and the Vasgra Cohort. Comparing diagnostic accuracy of 18F-FDG-PET/CT, contrast enhanced CT and combined imaging in patients with suspected vascular graft infections. Eur J Nucl Med Mol Imaging. 2019 Jun;46(6):1359-1368. doi: 10.1007/s00259-018-4205-y. Epub 2018 Nov 13. PMID 30426151
- [Derived] Anagnostopoulos A, Ledergerber B, Kuster SP, Scherrer AU, Naf B, Greiner MA, Rancic Z, Kobe A, Bettex D, Hasse B; VASGRA Cohort Study. Inadequate Perioperative Prophylaxis and Postsurgical Complications After Graft Implantation Are Important Risk Factors for Subsequent Vascular Graft Infections: Prospective Results From the Vascular Graft Infection Cohort Study. Clin Infect Dis. 2019 Aug 1;69(4):621-630. doi: 10.1093/cid/ciy956. PMID 30395220
- [Derived] Husmann L, Ledergerber B, Anagnostopoulos A, Stolzmann P, Sah BR, Burger IA, Pop R, Weber A, Mayer D, Rancic Z, Hasse B; VASGRA Cohort Study. The role of FDG PET/CT in therapy control of aortic graft infection. Eur J Nucl Med Mol Imaging. 2018 Oct;45(11):1987-1997. doi: 10.1007/s00259-018-4069-1. Epub 2018 Jun 11. PMID 29948106
- [Derived] Ajdler-Schaeffler E, Scherrer AU, Keller PM, Anagnostopoulos A, Hofmann M, Rancic Z, Zinkernagel AS, Bloemberg GV, Hasse BK; and the VASGRA Cohort. Increased Pathogen Identification in Vascular Graft Infections by the Combined Use of Tissue Cultures and 16S rRNA Gene Polymerase Chain Reaction. Front Med (Lausanne). 2018 Jun 4;5:169. doi: 10.3389/fmed.2018.00169. eCollection 2018. PMID 29915786
- [Derived] Husmann L, Sah BR, Scherrer A, Burger IA, Stolzmann P, Weber R, Rancic Z, Mayer D, Hasse B; VASGRA Cohort. (1)(8)F-FDG PET/CT for Therapy Control in Vascular Graft Infections: A First Feasibility Study. J Nucl Med. 2015 Jul;56(7):1024-9. doi: 10.2967/jnumed.115.156265. Epub 2015 May 14. PMID 25977463